CLINICAL TRIAL: NCT01497379
Title: Safety & Efficacy of Subretinal Implants for Partial Restoration of Vision in Blind Patients: A Prospective Mono- & Multicenter Clinical Study Based on Randomized Intra-individual Implant Activation in Degenerative Retinal Disease Patients.
Brief Title: Safety & Efficacy of Subretinal Implants for Partial Restoration of Vision in Blind Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Retina Implant AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: HKCTR-1198; RI-MC-CT-2009 (Registry Identifier: Clinicaltrials.gov)
Record Dates: First submitted 2011-12-15; First posted 2011-12-22 (Estimated); Last update posted 2017-03-29 (Actual); Status verified 2017-03

CONDITIONS: Retinal Degeneration; Retinitis Pigmentosa
Keywords: Hereditary retinal; degeneration outer; retinal layers; photoreceptor rods cones; Retinitis pigmentosa; blindness; reading ability; retina implant; subretinal
MeSH Terms: conditions — Retinal Degeneration; Retinitis Pigmentosa; Blindness | interventions — Retinaldehyde

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- intra-individual implant ON (Experimental): intra-individual implant activation
  Interventions: Procedure: surgical implantation of subretinal device
- intra-individual implant OFF (Placebo Comparator): intra-individual implant deactivation
  Interventions: Procedure: surgical implantation of subretinal device

INTERVENTIONS:
Procedure: surgical implantation of subretinal device — surgical implantation of subretinal device
  Other Names: Retinal implant, subretinal implant
  Arms: intra-individual implant ON
Procedure: surgical implantation of subretinal device — intra-individual implant OFF
  Other Names: Retinal implant, subretinal implant
  Arms: intra-individual implant OFF

SUMMARY:
Patients who are legally blind, caused by retinal degeneration of photoreceptor rods & cones (e.g. Retinitis pigmentosa), receive a subretinal implant to restore vision partially.

ELIGIBILITY:
Inclusion Criteria:

* Hereditary retinal degeneration of the outer retinal layers i.e. photoreceptor rods & cones.
* Pseudophakia
* Angiography shows retinal vessels adequately perfused, despite pathological RP condition.
* Age between 18 and 78 years.
* Blindness (at least monocular) i.e. visual functions not appropriate for localization of objects, self sustained navigation and orientation (impaired light localization or worse).
* Ability to read normal print in earlier life, optically corrected without magnifying glass.
* Willing and able to give written informed consent in accordance to EN ISO 14155 (section 6.7) and local legislation prior to participation in the study. Able to perform the study during the full time period of one year

Exclusion Criteria:

* Period of appropriate visual functions < 12 years / lifetime.
* Optical Coherence Tomography (OCT) shows significant retina edema &/or scar tissue within target region for implant.
* Retina detected as too thin to expect required rest-functionality of inner retina as shown via Optical Coherence Tomography (OCT).
* Lack of inner-retinal function, as determined by Electrically Evoked Phosphenes (EEP).
* Heavy clumped pigmentation at posterior pole
* Any other ophthalmologic disease with relevant effect upon visual function (e.g. glaucoma, optic neuropathies, trauma, diabetic retinopathy, retinal detachment).
* Amblyopia reported earlier in life on eye to be implanted
* Systemic diseases that might imply considerable risks with regard to the surgical interventions and anaesthesia (e.g. cardiovascular/ pulmonary diseases, severe metabolic diseases).
* Neurological and/or psychiatric diseases (e.g. M. Parkinson, epilepsy, depression).
* Hyperthyroidism or hypersensitivity to iodine
* Women who are pregnant or nursing, or women of childbearing potential who are not willing to use a medically acceptable means of birth control for the duration of the study, or women unwilling to perform a pregnancy test before entering the study.
* Participation in another interventional clinical trial within the past 30 days.

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2011-10; Primary Completion 2014-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Safety | 1 year
  treatment shows no permanent damage of function and structures that have been functional before surgery and no permanent damage to health and/or well being of patients
Efficacy | 1 year
  Activities of Daily Living & Mobility are significantly improved with implant-ON versus OFF, as shown via tests:
  * Activities of Daily Living tasks or
  * Recognition tasks or
  * Mobility or
  * a combination of the above

SECONDARY OUTCOMES:
Safety | 1 year
  Patient long term safety:
  * stability of implant function
  * stability of body structure & function related to implant system
Efficacy | 1 year
  Visual Acuity / Light-perception and/or Object-recognition are significantly improved with implant-ON versus OFF as shown via:
  * FrACT or
  * BaLM or
  * Grating test (e.g. BaGA) and/or Quality of life
  * Quality of life (questionnaire) or
  * a combination of the above

CONTACTS AND LOCATIONS:
Overall Officials: David Wong, Prof., MD, Principal Investigator — Chair Professor in Ophthalmology Eye Institute
Locations (1):
- Ophthalmology Eye Institute, University of Hong Kong, Hong Kong, Cyberport, Hong Kong

REFERENCES:
- [Result] Stingl K, Bartz-Schmidt KU, Besch D, Chee CK, Cottriall CL, Gekeler F, Groppe M, Jackson TL, MacLaren RE, Koitschev A, Kusnyerik A, Neffendorf J, Nemeth J, Naeem MA, Peters T, Ramsden JD, Sachs H, Simpson A, Singh MS, Wilhelm B, Wong D, Zrenner E. Subretinal Visual Implant Alpha IMS--Clinical trial interim report. Vision Res. 2015 Jun;111(Pt B):149-60. doi: 10.1016/j.visres.2015.03.001. Epub 2015 Mar 23. PMID 25812924
- See also: Hong Kong clinical trials registry — http://www.hkclinicaltrials.com/